CLINICAL TRIAL: NCT00587119
Title: Open-Label Pilot Study Evaluating Oral Budesonide in the Treatment of Patients With Primary Biliary Cirrhosis and Overlap Features of Autoimmune Hepatitis.
Brief Title: Oral Budesonide in the Treatment of Patients With Primary Biliary Cirrhosis and Overlap Features of Autoimmune Hepatitis
Acronym: PBC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr. Keith D. Lindor / PI, Mayo Clinic Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-003586; Budesonide
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Primary Biliary Cirrhosis; Autoimmune Hepatitis
Keywords: Urso; Budesonide; PBC; overlap AIH; PBC with overlap features of autoimmune hepatitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Hepatitis, Autoimmune | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single arm, active treatment
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Oral Budesonide, 3 mg three times daily, will be given for 1 year.
  Other Names: Entocort

SUMMARY:
The purpose of the study is to find out the effects Budesonide, 9 mg daily for one year, has on patients with Primary Biliary Cirrhosis with features of autoimmune hepatitis.

DETAILED DESCRIPTION:
Pilot Study of Budesonide for Primary Biliary Cirrhosis with overlap features of Autoimmune Hepatitis Primary biliary cirrhosis (PBC) is a chronic liver disease of unknown cause that may result in inflammation and destruction of the bile ducts inside the liver. Over time, cirrhosis and complications of liver failure may develop. Although treatment with ursodiol has been association with a reduction in liver enzymes (blood tests) and a reduction in the progression of the disease, some patients do not respond to ursodiol therapy. Patients with overlap features of Autoimmune Hepatitis (AIH) appear to be at higher risk of developing complications of disease even when on ursodiol. The purpose of this study is to evaluate the effects and safety of Budesonide in PBC with overlap features of AIH. Budesonide has unique effects on the immune system that may be helpful in the treatment of the disease.

Eligible participants will include those patients with a diagnosis of PBC with overlap features of AIH and in whom liver enzymes have not sufficiently improved with ursodiol therapy (the alkaline phosphatase is not less than twice upper normal). At entry all patients will have a history and physical examination, blood tests, bone densitometry and complete quality of life questionnaires. Patients will be prescribed Budesonide 9 mg to take daily for one year in addition to the ursodiol. The medication can be taken with or without food. Blood tests and symptoms diaries will be completed every 3 months. Patients will be contacted by phone to assess tolerance of the medication and any new health problems. At one year, patients will return for a history and physical and repeat blood tests and bone densitometry. Possible side-effects include bone mass loss (bone thinning), diarrhea, indigestion, nausea, joint pains, dizziness, headaches, weight gain and Cushing's syndrome. Other side-effects are possible. The medication and the tests will be billed to the patient or patient's insurance.

ELIGIBILITY:
Inclusion Criteria:

* Chronic cholestatic liver disease for greater than 6 months with alkaline phosphatase levels greater than 2 times the upper limit of normal.
* Positive AMA titer 1:40 or AMA > 1.0 U.
* Liver histology in the past (available for review) with features consistent with or diagnostic of PBC
* Ultrasound, computed tomography (CT), or cholangiography of the biliary tree which excludes biliary obstruction.
* The diagnosis of AIH necessary for evaluation of PBC-AIH overlap syndrome will be based on the revised International Autoimmune Hepatitis Group (IAHG) Scoring System.

Exclusion Criteria:

* Patients with other serious coexistent conditions such as pre-existing advanced malignancy or severe cardiopulmonary disease which would be expected to limit their expectancy to less than three years.
* Patients unable to provide informed consent.
* Treatment with methotrexate, corticosteroids, azathioprine, chlorambucil, cyclosporin, penicillamine, colchicine or chenodeoxycholic acid in the preceding three months.
* Anticipated need for transplantation in one year (Mayo survival model <80% one-year survival without transplant).
* Liver biopsy revealing stage IV disease.
* Evidence of portal hypertension such as esophageal varices, portal gastropathy, ascites or hepatic encephalopathy.
* Known history of portal vein thrombosis.
* Evidence of osteoporosis.
* Serum bilirubin >4 mg/dl.
* Age less than 21 years of age or greater than 75 years of age.
* Pregnancy.
* Breast-feeding.
* Active drug or alcohol use.
* Findings highly suggestive of liver disease of other etiology such as chronic alcoholic liver disease, chronic hepatitis B or C infection, hemochromatosis, Wilson's disease, 1-antitrypsin deficiency, non-alcoholic steatohepatitis or sclerosing cholangitis.
* Serum creatinine over 2.0 mg/dl.
* History of documented active peptic ulcer disease in preceding year.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
The main endpoint will be the percentage of patients with improvement in alkaline phosphatase to less than 1.5 times normal over one year and the percentage of patients with a reduction in their Mayo Risk Score over one year. | 1 year

SECONDARY OUTCOMES:
Effects of UDCA & budesonide on serum levels of alk phos, AST, total bilirubin, albumin, and prothrombin time, Mayo risk score and toxicity and tolerability of the budesonide/UDCA regimen, including effects on bone density. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Lindor, MD, Principal Investigator — Mayo Clinic